CLINICAL TRIAL: NCT05249894
Title: Evaluation of Infective Risk, Efficacy of Bacterial Prophylaxis and Validation of Sepsis Scores NEWS (National Early Warning Score) and qSOFA (Quick Sequential Organ Failure Assessment) in Patient With Acute Myeloid Leukemia Treated With Intensive Chemotherapy (LAM-SEPSIS)
Brief Title: Evaluation of Infective Risk, Efficacy of Bacterial Prophylaxis and Validation of Sepsis Scores NEWS (National Early Warning Score) and qSOFA (Quick Sequential Organ Failure Assessment) in Patient With Acute Myeloid Leukemia Treated With Intensive Chemotherapy
Acronym: LAM-SEPSIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Chiara Frairia, Medical Doctor in Hematology, A.O.U. Città della Salute e della Scienza
Other Study IDs: LAM-SEPSIS
Record Dates: First submitted 2022-01-20; First posted 2022-02-22 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Sepsis score; National Early Warning Score (NEWS); quick Sequential Organ Failure Assessment (qSOFA); chemotherapy-induced febrile neutropenia; Antibiotics prophylaxis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Chemotherapy-Induced Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of Infective Risk, Efficacy of Bacterial Prophylaxis and Validation of sepsis scores NEWS (National Early Warning Score) and qSOFA (Quick Sequential Organ Failure Assessment) in Patient With Acute Myeloid Leukemia Treated With Intensive Chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non M3 Acute Myeloid Leukemia according to WHO (World Health Organization) 2008 criteria
* Age >= 18 years and <= 70 years
* Patient had received intensive chemotherapy either as induction or consolidation regimen
* Period of observation: January 2001 - December 2019
* Written informed consent

Exclusion Criteria:

* Diagnosis of Acute Promyelocytic Leukemia (M3 AML)
* Age < 18 or >70 years
* Patient had not received intensive chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by Acute Myeloid Leukemia that had received between JAN2001 and DEC2019 an intensive chemotherapy cycle either as induction or consolidation regimen
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Mortality risk | At baseline (fever onset), change at 24 hours from baseline, change at 48 hours from baseline
  Ability of NEWS and qSOFA score to predict mortality risk calculating the area under the ROC (receiver operating characteristics) curve called AUROC (area under the ROC curve)

SECONDARY OUTCOMES:
Systemic Inflammatory Response Syndrome (SIRS) development | At baseline (fever onset), change at 24 hours from baseline, change at 48 hours from baseline
  Ability of NEWS and qSOFA score to predict SIRS development calculating the area under the ROC (receiver operating characteristics) curve called AUROC (area under the ROC curve)
Amine requirement | At baseline (fever onset), change at 24 hours from baseline, change at 48 hours from baseline
  Ability of NEWS and qSOFA score to predict vasoactive drugs requirement calculating the area under the ROC (receiver operating characteristics) curve called AUROC (area under the ROC curve)
Respiratory failure | At baseline (fever onset), change at 24 hours from baseline, change at 48 hours from baseline
  Ability of NEWS and qSOFA score to predict respiratory failure calculating the area under the ROC (receiver operating characteristics) curve called AUROC (area under the ROC curve)
Ventilation support | At baseline (fever onset), change at 24 hours from baseline, change at 48 hours from baseline
  Ability of NEWS and qSOFA score to predict ventilation support necessity calculating the area under the ROC (receiver operating characteristics) curve called AUROC (area under the ROC curve)
Intensive care unit (ICU) admission | At baseline (fever onset), change at 24 hours from baseline, change at 48 hours from baseline
  Ability of NEWS and qSOFA score to predict ICU admission calculating the area under the ROC (receiver operating characteristics) curve called AUROC (area under the ROC curve)
Bloodstream infections | From date of fever onset until the date of fever resolution, assessed up to 60 days
  Ability of NEWS and qSOFA score to predict severity of bloodstream infection calculating the area under the ROC (receiver operating characteristics) curve called AUROC (area under the ROC curve)
Number of infections | From date of neutrophils count <500/mmc until the day of neutrophils count >=500/mmc, assessed up to 60 days
  Cumulative incidence of infections in patients with levofloxacin prophylaxis vs. patients without levofloxacin prophylaxis

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy